CLINICAL TRIAL: NCT06957301
Title: Intrathecal Fentanyl and Dexmedetomidine Added to Bupivacaine for Subarachnoid Anaesthesia for Percutaneous Nephrolithotomy: A Randomized Superiority Trial
Brief Title: Intrathecal Fentanyl and Dexmedetomidine Added to Bupivacaine for Subarachnoid Anaesthesia for Percutaneous Nephrolithotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: serial number:0307226
Record Dates: First submitted 2025-04-12; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Percutaneous Nephrolithotomy (PCNL)
Keywords: percutaneous nephrolithotomy; intrathecal additive; dexametamodine; fentanyl

STUDY DESIGN:
Intervention Model Description: A randomized superiority trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group fentanyl (F) (Active Comparator): an injection of bupivacaine 0.5% (3.5 ml) + fentanyl 0.5 ml (25 μg) will be given intrathecal
  Interventions: Procedure: Intrathecal Fentanyl Group (F)
- Group dexmedetomidine( D) (Active Comparator): In Group dexmedetomidine( D), dexmedetomidine will be first diluted in normal saline to obtain a dose of 5 μg in 0.5 ml. Then, an injection of bupivacaine 0.5% (3.5 ml) + dexmedetomidine 0.5 ml (5 μg) will be administered intrathecally. Drug will be administered over 10 seconds (s) using 5 cc syringes with cephalad orientation of the spinal needle bevel.
  Interventions: Procedure: intrathecal dexmedetomidine group(D)

INTERVENTIONS:
Procedure: Intrathecal Fentanyl Group (F) — Group fentanyl (F), an injection of bupivacaine 0.5% (3.5 ml) + fentanyl 0.5 ml (25 μg) will be administered intrathecally.
  Arms: Group fentanyl (F)
Procedure: intrathecal dexmedetomidine group(D) — Group dexmedetomidine( D), dexmedetomidine will be first diluted in normal saline to obtain a dose of 5 μg in 0.5 ml. Then, an injection of bupivacaine 0.5% (3.5 ml) + dexmedetomidine 0.5 ml (5 μg) will be administered intrathecally. Drug will be administered over 10 seconds (s) using 5 cc syringes with cephalad orientation of the spinal needle bevel.
  Arms: Group dexmedetomidine( D)

SUMMARY:
Regular bupivacaine dosages are linked to considerable sympathetic block, as well as persistent and severe sensory and motor block, which may not be desired for certain individuals. Although diluted bupivacaine at low doses restricts the distribution of spinal block and produces a comparatively quick recovery, it might not offer a sufficient degree of sensory block.Bupivacaine's side effects and dosage requirements are lessened by the potentiating effects of the short-acting lipophilic opioid fentanyl and the more selective α2 agonist dexmedetomidine. These spinal adjuncts are used to extend analgesia in addition to lessening the negative effects of local anesthetics. According to a number of studies, when given intrathecally, α2 receptor agonists will increase the analgesia that subtherapeutic doses of local anesthetics like bupivacaine deliver because of their synergistic effects with little hemodynamic effects.The goal will be to determine if bupivacaine and fentanyl or bupivacaine and dexmedetomidine produced higher-quality anesthesia.

DETAILED DESCRIPTION:
Spinal anesthesia is a straightforward procedure that acts quickly. However, because of its neurotoxic effects, a common anesthetic like lidocaine has mostly been substituted by alternative substances like bupivacaine. Regular bupivacaine dosages are linked to considerable sympathetic block, as well as persistent and severe sensory and motor block, which may not be desired for certain individuals. Although diluted bupivacaine at low doses restricts the distribution of spinal block and produces a comparatively quick recovery, it might not offer a sufficient degree of sensory block. Bupivacaine's side effects and dosage requirements are lessened by the potentiating effects of the short-acting lipophilic opioid fentanyl and the more selective α2 agonist dexmedetomidine. These spinal adjuncts are used to extend analgesia in addition to lessening the negative effects of local anesthetics.

The danger of respiratory depression for lipophilic opioids, such as fentanyl and sufentanil, is primarily restricted to the first two hours following intrathecal injection. Because fentanyl is more lipid soluble than morphine, there is a significantly lower chance of delayed respiratory depression brought on by the rostral distribution of an intrathecal injected drug to respiratory centers.

Both visceral and somatic pain can be reduced by intrathecal α2 receptor agonists. Compared to clonidine (α2/α1 200:1), dexmedetomidine has greater selectivity for the α2 receptor (α2/α1 1600:1). According to a number of studies, when given intrathecally, α2 receptor agonists will increase the analgesia that subtherapeutic doses of local anesthetics like bupivacaine deliver because of their synergistic effects with little hemodynamic effects. The goal will be to determine if bupivacaine and fentanyl or bupivacaine and dexmedetomidine produced higher-quality anesthesia.

.

Objective:

The study's main goal is to evaluate patient satisfaction and sedation level. Comparing the two groups' analgesia duration, initial post-operative analgesia request, analgesia onset time (measured by pinpricking the T6 block level), peak block time, degree of motor blockade, and hemodynamic profiles will be the secondary outcome.

Methods and patients:

After obtaining Institutional Ethical Committee approval, this prospective randomised double-blinded study was carried out in a tertiary health care centre on 100 patients After obtaining Institutional Ethical Committee approval, this prospective randomised double-blinded study will be carried out in a tertiary health care centre on 100 patients of

Intervention:

Spinal anaesthesia will be performed in all patients in the sitting position. Under strict aseptic precautions, using 25G Quincke needle mid-line spinal puncture was performed at L2-L3 level.

In Group fentanyl (F), an injection of bupivacaine 0.5% (3.5 ml) + fentanyl 0.5 ml (25 μg) was administered intrathecally.

In Group dexmedetomidine( D), dexmedetomidine will be first diluted in normal saline to obtain a dose of 5 μg in 0.5 ml. Then, an injection of bupivacaine 0.5% (3.5 ml) + dexmedetomidine 0.5 ml (5 μg) will be administered intrathecally. Drug will be administered over 10 seconds (s) using 5 cc syringes with cephalad orientation of the spinal needle bevel. The patients were turned supine immediately after the injection of the drug.

Midazolame and fentanyle will be administered on request as rescue analgesic and for sedation if needed . post-operatively and side-effects such as hypotension, bradycardia, pruritus, vomiting, respiratory depression were also monitored. Pruritus was managed with i.v chlorpheniramine maleate.

ELIGIBILITY:
Inclusion Criteria:

* both sex aged between 18 and 60 years,
* belonging to American Society of Anaesthesiologists (ASA) physical status Grade I and II undergoing PCNL under spinal anaesthesia.

Exclusion Criteria:

* Patients with a history of spine surgery,
* infection at the injection site,
* coagulopathy,
* hypovolemia,
* increased intracranial pressure,
* indeterminate neurologic disease,
* spinal deformities,
* communication problems,
* known hypersensitivity to local anaesthetics, opioids or dexmedetomidine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
to evaluate patient satisfaction | at the end of the surgery (assessed up to 40 minutes)
  The level of patient's satisfaction was measured using five-point Likert scale ((1 = very dissatisfied, 2 = dissatisfied, 3 = neutral, 4 = satisfied, and 5 = very satisfied)
to evaluate the sedation grade | 10 minutes after giving the intervention , then after 30 minutes , then at the end of the surgery (assessed up to 40 minutes)
  5- Ramsay Sedation Score
  1. - Anxious, agitated/restless or both
  2. - Patient cooperative, oriented, and tranquil
  3. - Patient responds to commands only
  4. - Brisk response to a light glabellar tap or loud auditory stimulus
  5. - Sluggish response to light glabellar tap or loud auditory stimulus
  6. - Patient shows no response.

SECONDARY OUTCOMES:
to compare analgesia onset, duration ,peak sensory level | after giving the intervention every 1 minutes till reach level T6 (assessed up to 10 minutes)
  Sensory block level which will be defined as the loss of pain sensation to pin prick test in the midclavicular line, will be measured every1 min until it reached T6 level, and the surgeons will be asked to start. And record the time to reach peak sensory level .
to compare the initial post-operative analgesia request | 24 hour after surgery
  recording the time the patient need rescue analgesia post operative
to compare the degree of motor blockade between the two groups | at the time of peak sensory (up to 10 minutes) and then every 1hour for 3 hours post operative
  The degree of motor blockade at the time of peak sensory block and after end of surgery will be scored using a modified Bromage scale (MBS)(1)
  - (1) Complete motor block, (2) Almost complete motor block, patient is able to move only feet, (3) Partial motor block, patient is able to move the knees, (4) Detectable weakness of hip flexion, patient is able to raise the leg but is unable to keep it raised, (5) No detectable weakness of hip flexion, patient is able to keep the leg raised for 10s at least, (6) No weakness at all).
to compare the mean arterial blood pressure between the two groups | every 5 min up to 15 min after the intervention , then every 15 min during surgery and then for each hour after surgery in the ward(up to 4 hour).
  Mean blood pressure will be recorded every 5 min up to 15 min and then every 15 min during surgery then for each hour after surgery in the ward (up to 4 hour) .
  Hypotension, defined as mean BP less than 60 mm Hg will be treated by injection of ephedrine and crystalloids intravenous .
to record Post-operative and intraoperative complications | during the procedure ,24 hour postoperatively
  Post-operative and intraoperative complications (respiratory depression, vomiting ,nausea,pruitis)
to compare heart rate between to groups | every 5 min up to 15 min after the intervention , then every 15 min during surgery and then for each hour after surgery in the ward(up to 4 hour)
  Heart rate (HR) will be recorded every 5 min up to 15 min and then every 15 min during surgery then for each hour after surgery in the ward.
  Bradycardia was defined as HR <60 beats/min will be treated with intravenous atropine 0.3 mg increments.

CONTACTS AND LOCATIONS:
Overall Officials: Islam Elbardan, Dr, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of medicine ,Alexandria university, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No